CLINICAL TRIAL: NCT06529796
Title: A Phase 1, Open-label Study to Assess the Pharmacokinetics and Safety of a Single Dose of Inaxaplin in Subjects With Mild or Moderate Hepatic Impairment and in Matched Healthy Subjects
Brief Title: Evaluation of the Pharmacokinetics and Safety of Inaxaplin in Participants With Mild or Moderate Hepatic Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: VX20-147-006
Record Dates: First submitted 2024-07-26; First posted 2024-07-31 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Focal Segmental Glomerulosclerosis (FSGS)
MeSH Terms: conditions — Glomerulosclerosis, Focal Segmental

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1: Mild Hepatic Impairment (Experimental): Participants will receive a single dose of IXP on Day 1.
  Interventions: Drug: IXP
- Cohort 2: Matched Healthy Participants (Experimental): Healthy participants matched to Cohort 1 will receive a single dose of IXP on Day 1.
  Interventions: Drug: IXP
- Cohort 3: Moderate Hepatic Impairment (Experimental): Participants will receive a single dose of IXP on Day 1.
  Interventions: Drug: IXP
- Cohort 4: Matched Healthy Participants (Experimental): Healthy participants matched to Cohort 3 will receive a single dose of IXP on Day 1.
  Interventions: Drug: IXP

INTERVENTIONS:
Drug: IXP — Tablet for oral administration.
  Other Names: VX-147; Inaxaplin

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics, safety and tolerability of Inaxaplin (IXP) in participants with mild or moderate hepatic impairment and in matched healthy participants.

DETAILED DESCRIPTION:
This clinical trial information was submitted voluntarily under the applicable law and, therefore, certain submission deadlines may not apply. (That is, clinical trial information for this applicable clinical trial was submitted under section 402(j)(4)(A) of the Public Health Service Act and 42 CFR 11.60 and is not subject to the deadlines established by sections 402(j)(2) and (3) of the Public Health Service Act or 42 CFR 11.24 and 11.44.).

ELIGIBILITY:
Key Inclusion Criteria:

* Cohorts 1 and 3: Participants with Hepatic Impairment

  * Cohort 1 (mild impairment): defined as a Child-Pugh total score of 5 to 6 (Child-Pugh Class A)
  * Cohort 3 (moderate impairment): defined as a Child-Pugh total score of 7 to 9 (Child-Pugh Class B)
* Cohorts 2 and 4: Healthy Participants

  * Participants will be matched during screening to participants with mild (Cohort 1) or moderate (Cohort 3) hepatic impairment according to each of the following parameters: age (± 10 years); sex; and BMI (± 15%)

Key Exclusion Criteria:

* Cohorts 1 and 3: Participants with Hepatic Impairment

  * Acute febrile illness within 14 days and/or acute illness within 5 days before first dose of study drug
  * Participants who smoke
* Cohorts 2 and 4: Healthy Participants

  * Acute febrile illness within 14 days and/or acute illness within 5 days before first dose of study drug
  * Any condition possibly affecting drug absorption

Other protocol defined Inclusion/Exclusion criteria may apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2024-08-02 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of IXP | From Day 1 up to Day 10
Area Under the Concentration Versus Time Curve From the Time of Dosing Extrapolated to Infinity (AUC0-inf) of IXP | From Day 1 up to Day 10

SECONDARY OUTCOMES:
Safety and Tolerability as Assessed by Number of Participants With Adverse events (AEs) and Serious Adverse Events (SAEs) | From Day 1 up to Day 20

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Division of Clinical Pharmacology, University of Miami, Miami, Florida
  - GCP Research, St. Petersburg, Florida
  - Texas Liver Institute, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/independent-research/clinical-trial-data-sharing